## Document Cover Page

## **Study Title:**

Enhancing COVID-19 Vaccination Intentions by Eliciting Prosocial Altruistic Motives: Evaluating the Efficacy of a Brief Video-Based Intervention

NCT number: NCT04960228

**Date of Document:** May 7<sup>th</sup>, 2021



Centre intégré universitaire de santé et de services sociaux du Centre-Ouestde-l'Île-de-Montréal







## **Information and Consent Form**

**RESEARCH PROJECT:** Exploring changes in attitudes and beliefs related to the COVID-19 vaccine

This research study is funded by the McGill Interdisciplinary Initiative in Infection and Immunity (MI4).

## PRINCIPAL INVESTIGATOR

Dr Zeev Rosberger, PhD
 Lady Davis Institute for Medical Research - Jewish General Hospital
 & Department of Psychology - McGill University
 Institute of Community and Family Psychiatry
 4333, Côte Sainte-Catherine Road, Montreal, Qc, H3T 1E4

Would you prefer to complete the survey in English or French? Préférez-vous répondre à ce questionnaire en anglais ou en français ?

**English** 

Français

You are invited to complete this online survey to evaluate the impact of a brief video, or a brief informational text related to the COVID-19 pandemic. First, you will complete a brief survey about your attitudes, health behaviour and intentions, and you will then be randomly assigned to

one of two conditions 1) to watch a brief video or 2) to read a brief informational text. After this, you will be asked a few more questions concerning your reactions to the video or the text. The information you give us will be extremely helpful in deciding how to educate the Canadian population about preventing COVID-19 virus transmission, hospitalizations, and deaths. You can refuse to answer any question in the survey.

We recommend having a strong and stable Internet connection while you complete the survey.

This survey should take approximately 10 minutes to complete. Your participation in this study is voluntary. You are free to choose whether or not to participate. You can withdraw from the study at any time and for any reason. If you withdraw from this research study before it ends, the information we already collected from you will be kept. You will be compensated approximately \$2.50-\$3 for this study depending on how you choose to use your rewards.

You may be contacted again at some point in the next few months, for another survey part of the same research project. Should this be the case, your participation to this second survey would once again be entirely voluntary.

All the information collected in the context of this research project will remain confidential. Your information will be collected anonymously. This data will be held on a secure password-protected file share on the server at the Lady Davis Institute for Medical Research, at the CIUSSS West-Central Montreal for 10 years. Principal Investigator Dr Zeev Rosberger is responsible for the data. By responding to this online survey, your identity will not be known. Results may be published in specialized journals, be presented in conferences, or be discussed in knowledge exchange activities, but it will be impossible to identify you. Dynata only uses identifying socio-demographic information to recruit eligible participants according to our study's criteria. However, none of this information is communicated to the research team. Dynata will send anonymous survey data to the research team.

You will not receive any direct personal benefit from participating in this study, but we hope that the research results will contribute to educating the population about preventing COVID-19 virus transmission, hospitalizations, and deaths.

Participating in this research study has no known or serious risks. However, it is possible that some of the information contained in the survey may cause you to experience discomfort or upset. If you feel any discomfort, you are free to stop at any time or refuse to answer any question.

If you do experience any discomfort as the result of completing the survey, you can get access to mental health support in your area through the resources available on the government web page: https://www.canada.ca/en/public-health/services/mental-health-services/mental-health-get-help.html.

For additional information on the COVID-19 vaccines, you can visit the websites indicated at the end of the survey.

In addition, if you have any questions regarding this research study, you can contact the principal investigator, Dr Zeev Rosberger at 514 340-8222 ext 24215 or at zeev.rosberger@mcgill.ca or the study coordinator, Gabrielle Griffin-Mathieu, at 514 340-8222 ext 23978 or at gabrielle.griffin@ladydavis.ca.

For all questions concerning your rights during your participation in this study, or if you have any complaints or comments regarding your experience in taking part in this research study, you can contact the Local Commissioner of Complaints and Quality of Service of the CIUSSS du Centre-Ouest-de-l'Île-de-Montréal or the ombudsman of the institution at (514) 340-8222, ex. 24222.

By completing this survey, you consent to be part of this study.